CLINICAL TRIAL: NCT00420628
Title: A Safety and Efficacy Study of Zylet® (Loteprednol Etabonate 0.5% and Tobramycin 0.3% Ophthalmic Suspension) Compared to Vehicle in the Management of Lid Inflammation (Chalazion/Hordeolum) in Pediatric Subjects
Brief Title: Pediatric Zylet Safety and Efficacy Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 459
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-09

CONDITIONS: Chalazion; Hordeolum
MeSH Terms: conditions — Chalazion; Hordeolum | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol/Tobramycin (Experimental): 0.5% loteprednol etabonate with 0.3% tobramycin opthalmic suspension
  Interventions: Drug: loteprednol etabonate/tobramycin opthalmic suspension
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: vehicle

INTERVENTIONS:
Drug: loteprednol etabonate/tobramycin opthalmic suspension — Topical ophthalmic drug: 0.5% loteprednol etabonate with 0.3% tobramycin 4 times a day (QID) days 1-7, 2 times a day (BID) days 8-14. Warm compresses were applied to affected eyes 2 times a day prior to application of study medication.
  Other Names: Zylet
  Arms: Loteprednol/Tobramycin
Drug: vehicle — topical ophthalmic vehicle was applied 4 times a day (QID) days 1-7, 2 times a day (BID) days 8-14. Warm compresses were applied to affected eyes 2 times a day prior to application of study medication.
  Arms: Vehicle

SUMMARY:
A multicenter study to evaluate the safety and efficacy of Zylet compared to vehicle in children aged 0-6 for the management of lid inflammation (chalazion/hordeolum)

ELIGIBILITY:
Inclusion Criteria:

* Child, 0 to 6 years of age, any sex and race
* Subject must have a clinical diagnosis of lid inflammation (e.g. Chalazion/Hordeolum) in at least one eye. If both eyes are diagnosed with lid inflammation, both eyes will be treated
* In good health (no current or past relevant medical history), based on the judgment of the investigator
* Parent/guardian is able and willing to follow instructions and provide informed consent

Exclusion Criteria:

* Known hypersensitivity to corticosteroids, loteprednol etabonate, or any component of the study medication
* Known hypersensitivity to aminoglycosides, tobramycin, or any component of the study medication
* Use of concurrent ocular therapy with non-steroidal anti-inflammatory agent (NSAID), mast cell stabilizer, antihistamine, or decongestant within 48 hours before and during the study
* Use of oral or topical ophthalmic corticosteroids (other than study medication) within 48 hours before and during the study
* Use of systemic antibiotics within 72 hours before and during the 14 day study medication treatment duration
* Use of topical ophthalmic antibiotics (other than the study medication) within 72 hours before and during the study
* History of ocular surgery, including laser procedures, within the past six months
* Anticipation that surgical intervention for lid inflammation will be required prior to completion of the study
* Subjects with suspected vernal conjunctivitis, glaucoma of any kind, viral or bacterial conjunctivitis, preseptal cellulitis requiring systemic antibiotics, dacryocystitis, uveitis, or any other disease conditions that could interfere with the safety and efficacy evaluations of the study medication
* History of any severe/serious ocular pathology or medical condition that could result in the subject's inability to complete the study
* Participation in an ophthalmic drug or device research study within 30 days prior to entry in this study
* Unlikely to comply with the protocol instructions for any reason

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Comstock, OD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Pediatric Ophthalmology of Erie, Erie, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 108 subjects aged 0-6 years with lid inflammation were recruited from 15 clinic locations in the US. First subject was enrolled on 11/07/2006, last subject visit was 1/5/2009.
Pre-assignment Details: 108 subjects were randomized to receive loteprednol/tobramycin or its vehicle in a 2:1 ratio. Subjects will receive warm compress lid treatment 2 times daily, before administration of study medication (as applicable) for the 14-day treatment duration.
Groups:
- Loteprednol/Tobramycin: 0.5% loteprednol etabonate with 0.3% tobramycin opthalmic suspension administered into affected eye(s) for 14 days
- Vehicle: Vehicle used in the study drug administered into affected eye(s) for 14 days
Period: Overall Study
Arm/Group | Loteprednol/Tobramycin | Vehicle
Started | 72 | 36
Completed | 63 | 32
Not Completed | 9 | 4
Not completed — Withdrawn by parent or gaurdian | 5 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol/Tobramycin | Vehicle | Total
Number analyzed (Participants) | 72 | 36 | 108
Age, Customized [Number; unit: participants]
  Age 0-6 years | 72 | 36 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 23 | 60
  Male | 35 | 13 | 48
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 1 | 4
  Black or African American | 10 | 7 | 17
  White | 52 | 25 | 77
  Other | 7 | 3 | 10

OUTCOME MEASURES:

1. Secondary Outcome: Investigators Global Assessment of the Clinical Condition
Description: The efficacy endpoints for this study consisted of reduction of inflammation as measured by the IGA of the clinical condition. Changes in clinical condition measured as improved, unchanged or worsened.
Time Frame: Visit 3, day 8
Population: Efficacy Sample, subjects with non-missing data. Day 15 (Visit 3)
Measure: Number; unit: Participants
Arm/Group | Loteprednol/Tobramycin | Vehicle
Number analyzed (Participants) | 63 | 32
Participants
  Improved | 36 [44.0 to 69.5] | 17 [34.7 to 70.9]
  Unchanged | 25 | 13
  Worse | 2 | 2

2. Primary Outcome: Treatment Emergent Adverse Events
Description: Study eye - Safety Population, At all visits 1,2,3
Time Frame: day 1, day 8, day 15
Population: Safety population, Study eye
Measure: Number; unit: participants
Arm/Group | Loteprednol/Tobramycin | Vehicle
Number analyzed (Participants) | 72 | 36
participants
  Conjunctivitis | 2 | 0
  Meibomianitis | 1 | 1
  Eyelid edema | 0 | 1

3. Secondary Outcome: Assessment of Ocular Signs in the Study Eye - Visit 1
Description: Lid edema, lid erythema, palpebral conjunctival injection, meibomium plugging measured on a scale of 0-4 none, minimal, mild, moderate, severe.
Time Frame: Visit 1 (day 1)
Population: Efficacy sample, non-missing data
Measure: Mean (Standard Deviation); unit: Units on a scale 0-4
Arm/Group | Loteprednol/Tobramycin | Vehicle
Number analyzed (Participants) | 66 | 34
Units on a scale 0-4
  Lid Edema | 1.97 (0.84) | 2.06 (0.95)
  Lid Erythema | 1.98 (1.10) | 1.82 (1.22)
  Palpebral Conjunctival Injection | 1.85 (1.13) | 1.79 (0.98)
  Meibomian Plugging | 1.44 (1.04) | 1.59 (1.26)

4. Secondary Outcome: Assessment of Ocular Signs in the Study Eye - Visit 2
Description: as for outcome 3
Time Frame: Visit 2 (day 8)
Population: Efficacy population - Study eye
Measure: Mean (Standard Deviation); unit: Units on a scale 0-4
Arm/Group | Loteprednol/Tobramycin | Vehicle
Number analyzed (Participants) | 66 | 32
Units on a scale 0-4
  Lid Edema | 1.47 (0.92) | 1.38 (0.94)
  Lid Erythema | 1.41 (1.01) | 1.47 (1.08)
  Palpebral Conjunctival Injection | 1.41 (1.01) | 1.16 (0.92)
  Meibomian Plugging | 1.06 (1.02) | 1.00 (1.11)

5. Secondary Outcome: Assessment of Ocular Signs in the Study Eye - Visit 3
Description: as for outcome 3
Time Frame: Visit 3 (day 15)
Population: Efficacy sample - Study eye
Measure: Mean (Standard Deviation); unit: Units on a scale 0-4
Arm/Group | Loteprednol/Tobramycin | Vehicle
Number analyzed (Participants) | 63 | 32
Units on a scale 0-4
  Lid Edema | 1.03 (0.90) | 1.41 (1.10)
  Lid Erythema | 1.00 (0.88) | 1.50 (1.14)
  Palpebral Conjunctival Injection | 1.11 (0.95) | 1.09 (1.09)
  Meibomian Plugging | 0.86 (1.12) | 1.16 (1.22)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Loteprednol/Tobramycin | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/36
Other Adverse Events (participants affected / at risk) | 0/72 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol/Tobramycin (N=72) | Vehicle (N=36)
bilateral subdural hematoma (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the investigator(s) after the review by, and in consultation and agreement with Bausch & Lomb, and such that confidential or proprietary information is not disclosed.

Prior to publication or presentation, a copy of the final text should be forwarded by the investigator(s) to Bausch & Lomb or its designee, for comment.